CLINICAL TRIAL: NCT06354478
Title: A Randomized, Double-blind Study to Compare the Efficacy of Intravenous Dexmedetomidine Infusion, Oral Gabapentin and Their Combination on Postoperative Analgesia in Cancer Patients Undergoing Modified Radical Mastectomy
Brief Title: IV Dexmedetomidine vs Oral Gabapentin and Their Combination for Postoperative Analgesia in Cancer Patients Undergoing Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ms-103-2021
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Pain, Postoperative; Pain, Acute
Keywords: Breast Cancer; Perioperative pain; Dexmedetomidine; Gabapentin
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Acute Pain | interventions — Dexmedetomidine; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both patients and Investigator for postoperative pain will be blinded:
  * Group 1(D): (n=30) Patients will receive oral placebo starch capsules 1 hour preoperatively and intraoperative intravenous infusion of dexmedetomidine with general anaesthesia.
  * Group 2(G): (n=30) Patients will receive oral gabapentin capsules for 1 hour preoperatively and intraoperative intravenous saline infusion with general anaesthesia.
  * Group 3(DG): (n=30) Patients will receive oral gabapentin capsules for 1 hour preoperatively and intraoperative intravenous infusion of dexmedetomidine with general anaesthesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- D group (Experimental): D group: Patients will receive two oral placebo capsules (starch capsules) 1 hour before surgery, and then will receive a loading dose of 1µg/kg of dexmedetomidine made to 50 ml using normal saline and given intravenously just before induction of anaesthesia over 10 minutes while patient vital signs monitored followed by intravenous infusion of dexmedetomidine diluted in normal saline with a dose of 0.5µg/kg/hour starts with induction of anaesthesia at a rate of 10 ml/hour through identical syringe pump until skin closure.
  Interventions: Drug: Dexmedetomidine Hydrochloride 0.5 MG/ML
- G group (Experimental): G group: Patients will receive two oral gabapentin (300 mg) capsules for a total of 600 mg gabapentin (Neurontin; Pfizer, Cairo, Egypt) 1 hour before surgery, and then will receive 50 ml of normal saline given intravenously just before induction of anaesthesia over 10 minutes while patient vital signs monitored followed by intravenous normal saline infusion intraoperatively starts with induction of anaesthesia at a rate of 10 ml/hour through identical syringe pump until skin closure.
  Interventions: Drug: Gabapentin
- DG group (Experimental): DG group: Patients will receive two gabapentin (300 mg) capsules for a total of 600 mg gabapentin 1 hour before surgery, and then will receive a loading dose of 1µg/kg of dexmedetomidine made to 50 ml using normal saline and given intravenously just before induction of anaesthesia over 10 minutes while patient vital signs monitored followed by intravenous infusion of dexmedetomidine diluted in normal saline with a dose of 0.5µg/kg/hour starts with induction of anaesthesia at a rate of 10 ml/hour through identical syringe pump until skin closure.
  Interventions: Drug: Dexmedetomidine Hydrochloride 0.5 MG/ML; Drug: Gabapentin

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride 0.5 MG/ML — Will be used either alone or in combination of gabapentin
  Arms: D group; DG group
Drug: Gabapentin — Will be used either alone or in combination of Dexmedetomidine
  Arms: DG group; G group

SUMMARY:
Breast cancer is the most common malignant tumour among females with an incidence of about 2.1 million women every year.Nearly about 40-60% of breast surgery patients develop severe acute postoperative pain.⁴ Opioids are the current best standard drugs for postoperative pain relief, however, exposure to large doses of opioids leads to multiple side effects like prolonged sedation, respiratory depression, nausea, and vomiting.We are comparing two different drugs and their combination for perioperative analgesia for MRM.

This work is a comparative study that aims to compare the analgesic effects of perioperative IV infusion of dexmedetomidine, preoperative oral gabapentin, and their combination in patients undergoing modified radical mastectomy surgery regarding the time of first rescue analgesia, postoperative morphine consumption, and possible complications.

DETAILED DESCRIPTION:
Introduction:

Breast cancer is the most common malignant tumour among females with an incidence of about 2.1 million women every year. It is the greatest cancer-related mortality among women approximately 15% of all cancer mortality. In addition to that, Egypt follows the international incidence with breast cancer being the most common malignancy among females with 18,660 patients each year.¹ Modified Radical Mastectomy (MRM) is one of the main surgical treatments of breast cancer. Accordingly, it is an account for 31% of all breast surgery cases.² The common modality for anaesthesia for MRM is general anaesthesia with or without regional blocks.³

Nearly about 40-60% of breast surgery patients develop severe acute postoperative pain.⁴ Opioids are the current best standard drugs for postoperative pain relief, however, exposure to large doses of opioids leads to multiple side effects like prolonged sedation, respiratory depression, nausea, and vomiting.⁵ Moreover, the use of opioids inhibits cell-mediated immunity with an increase in tumour angiogenesis, cell migration, and metastasis in addition to the progression of the cell cycle. Therefore, plans other than opioids are recommended without losing proper and effective analgesia, especially in breast cancer patients who are more sensitive to develop opioid tolerance and addiction.⁶ So it became a necessity to find safe analgesic techniques for these patients by using different techniques like adjuvant therapies or multimodal analgesia by combining different drugs with different mechanisms of action together to increase the quality of postoperative analgesia and to decrease the need for high doses of systemic opioids and their related side addiction.⁷'⁸

Alpha-2 agonists including clonidine and dexmedetomidine have been used perioperatively. Dexmedetomidine is different from clonidine in two properties. It has more affinity for the alpha-2 receptor (8 times that of clonidine) and is easier to titrate.⁹ Also, dexmedetomidine is a highly selective alpha-2 adrenergic receptor agonist that has sedative, analgesic, anaesthetic-sparing properties without causing any respiratory depression.¹⁰ Dexmedetomidine can be a good anaesthetic premedication because of its sympatholytic effect to attenuate the sympathetic stress response to perioperative stresses like laryngoscopy and intubation.¹¹ The analgesic effect provided by dexmedetomidine is mediated mainly through interaction at alpha-2a within the spinal cord, where drug activity attenuates nociceptive signal transduction. And although dexmedetomidine when given alone has been documented to reduce pain, it has a synergistic or additive effect when combined with opioids.¹²

Another promising drug for postoperative pain management is gabapentin. It binds to the α-2 δ subunit of voltage-gated calcium channels and preventing the release of nociceptive neurotransmitters like glutamate, substance P, and noradrenaline.¹³ Evidence suggests that, in addition to its effectiveness as an analgesic for patients with neuropathic pain and chronic pain syndromes, gabapentin also provides effective postoperative analgesia when given before an operation.¹⁴'¹⁵ Therefore the combination of IV dexmedetomidine and oral gabapentin due to their analgesic effects would be more effective in reducing postoperative analgesic consumption and providing prolonged postoperative analgesia after a modified radical mastectomy.

To the best of researchers' knowledge, comparing the effect of perioperative intravenous dexmedetomidine infusion, preoperative oral gabapentin and their combination on the total consumption of intraoperative and postoperative opioids in patients undergoing modified radical mastectomy was not investigated before.

Aim of the work:

This work is a comparative study that aims to compare the analgesic effects of perioperative IV infusion of dexmedetomidine, preoperative oral gabapentin, and their combination in patients undergoing modified radical mastectomy surgery regarding the time of first rescue analgesia, postoperative morphine consumption, and possible complications.

Objectives:

To assess the analgesic outcomes of perioperative IV infusion of dexmedetomidine, preoperative oral gabapentin and their combination in controlling acute postoperative pain in modified radical mastectomy regarding:

* The time of first rescue analgesia during the first 24 hours postoperatively.
* Intraoperative fentanyl consumption.
* Postoperative morphine consumption.
* Postoperative VAS scores.
* Intra & postoperative complications of study drugs.

Hypothesis:

We assume that the combination of preoperative oral gabapentin and intraoperative IV dexmedetomidine infusion can provide more analgesic effect than either drug alone in the form of delaying first rescue analgesia time, reducing the total amount of opioid consumption, and improving postoperative VAS score.

Ethical Considerations:

This study will be conducted after the approval of the research committee of the department of anaesthesia, surgical ICU, and pain management in Kasr Alainy Hospital, Cairo University, and the ethical committee of the Faculty Of Medicine, Cairo University. Informed consent will be taken from all patients included in the study.

Methodology:

Patients will be assessed the day before surgery in a preoperative visit for evaluating their medical status, laboratory investigations, and for fulfilling all the above inclusion and exclusion criteria. The patients will be instructed how to report pain using the visual analogue scale (VAS) score rating, in which 0 = "no pain" and 10 = "worst possible pain. All groups of the study will be premedicated with I.V 0.02 mg/kg midazolam 30 minutes preoperatively. Heart rate (HR), mean arterial blood pressure (MBP) will be monitored before the induction of anaesthesia (baseline values), immediately before surgical incision, and at 15 min intervals intraoperatively. Also, the patients will be randomly assigned into three equal comparable groups, each of which 30 patients, using computer-generated random numbers.

D group: Patients will receive two oral placebo capsules (starch capsules) 1 hour before surgery, and then will receive a loading dose of 1µg/kg of dexmedetomidine made to 50 ml using normal saline and given intravenously just before induction of anaesthesia over 10 minutes while patient vital signs monitored followed by intravenous infusion of dexmedetomidine diluted in normal saline with a dose of 0.5µg/kg/hour starts with induction of anaesthesia at a rate of 10 ml/hour through identical syringe pump until skin closure.

G group: Patients will receive two oral gabapentin (300 mg) capsules for a total of 600 mg gabapentin (Neurontin; Pfizer, Cairo, Egypt) 1 hour before surgery, and then will receive 50 ml of normal saline given intravenously just before induction of anaesthesia over 10 minutes while patient vital signs monitored followed by intravenous normal saline infusion intraoperatively starts with induction of anaesthesia at a rate of 10 ml/hour through identical syringe pump until skin closure.

DG group: Patients will receive two gabapentin (300 mg) capsules for a total of 600 mg gabapentin 1 hour before surgery, and then will receive a loading dose of 1µg/kg of dexmedetomidine made to 50 ml using normal saline and given intravenously just before induction of anaesthesia over 10 minutes while patient vital signs monitored followed by intravenous infusion of dexmedetomidine diluted in normal saline with a dose of 0.5µg/kg/hour starts with induction of anaesthesia at a rate of 10 ml/hour through identical syringe pump until skin closure.

Dexmedetomidine or saline infusion loading started 10 minutes before the induction of anaesthesia while patient vital signs monitored, and Maintenance started with induction of anaesthesia and continued until skin closure at the end of surgery.

This study is a double-blind study, so neither the participants nor the experimenters will know who is receiving a particular treatment. The drugs will be prepared by an anaesthesiologist who has no further role in the study, the doses of administered IV drugs will be calculated according to the patient's body weight and they will be supplied as two syringes labelled respectively as: ( loading ) syringes which will contain 50 ml of normal saline or a loading dose of dexmedetomidine made to 50 ml using normal saline and both will be given intravenously over 10 minutes just before induction of anaesthesia while patient vital signs monitored and ( Maintenance ) syringes that will contain normal saline or a maintenance dose of dexmedetomidine diluted in normal saline and both will be given intravenously with the induction of anaesthesia at a rate of 10 ml/hour and continued until skin closure. All syringes pump will be used in the study will be identical. In addition to this, both placebo capsules (starch capsules) and gabapentin capsules (Neurontin 300mg) will be identical-looking capsules yellow in colour and capsule in shape. Also, the surgical team, the patients, the anaesthesiologists, and the investigators responsible for collecting intraoperative and postoperative recorded data did not know about the groups' allocation.

3. Anaesthesia Management:

The patients included in the study will be kept fasting for at least six hours before surgery and will be monitored continuously using electrocardiography, non-invasive blood pressure, peripheral oxygen saturation, and end-tidal carbon dioxide - using the Datex-Ohmeda S5 anaesthesia monitor, model no: USE1913A - throughout the surgical procedure. The intravenous (IV) access will be secured using a 20 gauge (G) cannula for IV fluid management and another IV access for the infusion of the study drugs.

Induction of general anaesthesia in all study groups will be performed using a regimen of IV 2 μcg/kg fentanyl and propofol IV 2 mg /kg. Tracheal intubation will be facilitated using 0.5 mg/kg IV of Atracurium. Anaesthesia will be maintained with inhaled sevoflurane in oxygen-enriched air (FiO 2=0.5) and top-up doses of atracurium (0.1 mg/kg ) IV will be administered as required guided by a nerve stimulator. All patients will be mechanically ventilated aiming to keep end-tidal carbon dioxide within the range of 30-35 mmHg. All patients will receive 1 g of IV paracetamol. The total intraoperative fentanyl consumption will be recorded in all study groups. Bispectral index (BIS) will be used for monitoring the depth of anaesthesia, with target BIS values from 40 to 60, because all the study drugs have a synergistic effect with inhaled anaesthesia.

Ringer acetate will be infused to replace any fluid deficit, maintenance, and losses. Hypotension will be defined as MBP less than 60mmHg or less than 70% from baseline. episodes of hypotension will be treated with ringer acetate boluses and/or 5mg ephedrine in incremental doses to maintain mean blood pressure above 70 mmHg. Additional bolus doses of fentanyl 0.5µg/kg will be given if the mean blood pressure or heart rate rises above 20% of baseline values.

At the end of the surgery, the residual neuromuscular blockade will be reversed using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg), and extubation will be performed after complete recovery of the airway reflexes. The patients will be transferred to the post-anaesthesia care unit then according to the modified Aldrete discharge scale, the patients will be shifted to the ward when the patient achieves an Aldrete score of 9/10.¹⁶ MBP, heart rate, and VAS pain score will be noted immediately on arrival in the post-anaesthesia care unit and at 2, 6, 12, 18, and 24 h postoperatively. All patients will be given paracetamol postoperatively 1 g IV every 8 hours until discharged. Rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the pain score was >3 with a maximum allowed daily dose of 0.5 mg/kg/24 hours. The time of the first rescue analgesia and the total amount of morphine given in the first 24 hours postoperatively will be recorded in the three groups.

Side effects such as nausea, vomiting, sedation, hallucination, respiratory depression (respiratory rate <10/min.), Postoperative nausea and vomiting (PONV) as side effects of morphine will be recorded upon arrival to PACU and at 2, 6, 12, 18, and 24 h postoperatively on a four-point verbal scale¹⁷ : (none =no nausea, mild = nausea but no vomiting, moderate = vomiting one attack, severe = vomiting >one attack). 0.1 mg/kg of IV ondansetron will be given to patients with moderate or severe postoperative nausea and vomiting.

Sedation will be assessed and scored at the same times of assessment of VAS of pain at 2, 6, 12, 18, and 24 h postoperatively and in the recovery room with Ramsay scores¹⁸ : (1 = anxious or restless or both; 2 = cooperative, orientated, and tranquil; 3 = responding to commands; 4 = brisk response to a stimulus; 5 = sluggish response to a stimulus, and 6 = no response to stimulus) excessively high Sedation level with Ramsay 5 or 6, adequate sedation levels needing observation with Ramsay 2 to 4 and inadequate or insufficient sedation level with Ramsay 1.

Statistical Methods:

Sample size justification:

The aim of this study is to compare the analgesic effects of perioperative IV infusion of dexmedetomidine and preoperative oral gabapentin in patients undergoing modified radical mastectomy surgery. Based on the previous work by (Grover et al., 2009)¹⁹, who reported the mean duration time of first rescue analgesia was 90±61.1 minutes and (Alzeftawy & Elsheikh 2015)²⁰ who reported 125 ± 25.7 minutes for Dexmedetomidine infusion. Using power 80% and 5% significance level; 30 patients in every group will be required. The sample size is calculated using G*Power program²¹ (University of Düsseldorf, Düsseldorf, Germany).

Statistical analysis:

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 24 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Data will be explored for normality using Kolmogrov-Smirnov test and Shapiro-Wilk test. Comparisons between 3 groups for normally distributed numeric variables will be done using the ANOVA while for non normally distributed numeric variables will be done by Kruskal Wallis test. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

Categorical data will be described as numbers and percentages and comparisons will be done by chi square test or fisher exact as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* ● Female physical status ASA I, II.

  * Body mass index (BMI): 20 kg/m2- 40 kg/m2.
  * A patient undergoing modified radical mastectomy under general anaesthesia.

Exclusion Criteria:

* ● Patient refusal.

  * Known sensitivity or contraindication to study drugs (e.g.: dexmedetomidine, gabapentin, or morphine ).
  * History of psychological disorders, chronic pain, and/or sympathetic disorders.
  * Patients receiving medications that are considered to result in tolerance to opioids as those who are receiving medications for cancer pain (e.g. tramadol and hydromorphone).
  * Significant liver insufficiency (liver enzymes more than two folds or severe liver cirrhosis) or renal insufficiency (plasma creatinine more than 1.5 mg/dl).
  * Severe respiratory disorders (e.g. Chronic obstructive pulmonary disease, Bronchial asthma), or cardiac disorders (e.g. ischemic heart disease, regional motion wall abnormality, EF< 50%).
  * Pregnancy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
The time to first rescue analgesia during the first 24 hour Postoperatively. | 24 hrs
  Time from postoperative recovery till the patients have pain enough requesting analgesia

SECONDARY OUTCOMES:
Total postoperative morphine consumption till the first 24 hours | 24 hrs
  total dose of morphine received
The degree of postoperative sedation according to Ramsay scores | 2 hrs
  postoperative level of sedation
VAS scores both at rest and during shoulder movement | 24 hrs
  scoring of pain intensity 0-10
Postoperative nausea and vomiting (PONV) as side effects of morphine. | 24 hrs
  will be classified to none-mild-moderate-severe

CONTACTS AND LOCATIONS:
Overall Officials: Ashgan Raouf Ali, Professor, Study Chair — Anaesthesiology Faculty of Medicine - Cairo University; Heba Ismail Ahmed Nagy, Professor, Study Director — Anaesthesiology Faculty of Medicine - Cairo University; Mina Samir Said Khalil, Principal Investigator — Anaesthesiology National Cancer Institute - Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No